CLINICAL TRIAL: NCT00031369
Title: In Vivo Mapping Of Structural and Biochemical Abnormalities In Patients With Primary Focal Dystonia
Brief Title: Brain Anatomy in Dystonia
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020132; 02-N-0132
Record Dates: First submitted 2002-03-02; First posted 2002-03-04 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-03-10

CONDITIONS: Dystonia; Healthy
Keywords: MRI; Writer's Cramp; Movement Disorder; Gray Matter; Brain Morphology; Dystonia; Focal Hand Dystonia; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Dystonia; Dystonic Disorders; Movement Disorders; Dystonia, Focal, Task-Specific

SUMMARY:
This study will use high-resolution magnetic resonance imaging (MRI) to look for subtle differences in brain anatomy between patients with focal hand dystonia (also called writer s cramp) and healthy normal volunteers. Patients with hand dystonia have prolonged muscle contractions that cause sustained twisting movements and abnormal postures. These abnormal movements often occur with activities such as writing, typing, playing certain musical instruments such as guitar or piano, or playing golf or darts.

Patients with focal hand dystonia and healthy volunteers will be enrolled in this study. Patients will be recruited from NINDS s database of patients with focal hand dystonia. Volunteers will be selected to match the patients in age, sex and handedness.

This study involves two visits to the NIH Clinical Center. The first visit is a screening visit, in which patients and volunteers will have a medical history, physical examination, neurological examination, and assessment of handedness. Women of childbearing age will be screened with a pregnancy test. Pregnant women are exclude from this study.

Those who join the study will return for a second visit for magnetic resonance imaging. MRI uses a magnetic field and radio waves to produce images of the brain. For the procedure, the participant lies still on a stretcher that is moved into the scanner (a narrow cylinder containing the magnet). Earplugs are worn to muffle loud noises caused by electrical switching of radio frequency circuits used in the scanning process. The scan will last about 45 to 60 minutes, at most. Some volunteers may be asked to return for a third visit to obtain a second MRI on a different scanner.

DETAILED DESCRIPTION:
Objective

The term, dystonia, is used to describe a syndrome characterized by prolonged muscle contractions causing sustained twisting movements and abnormal postures of the affected body part(s). Although no structural brain abnormalities have been definitively demonstrated in the visual inspection of MRI scans from patients with primary focal dystonia, there are several lines of evidence for subtle structural brain abnormalities at both the subcortical and cortical levels. We hypothesize that those abnormalities might be detected by using appropriate acquisition and analysis methods.

Study population

This research will be conducted using patients with primary focal dystonia and normal volunteers.

Design

By using high-resolution 3D structural magnetic resonance imaging (MRI) of the brain and voxel-based morphometry (VBM), and diffusion tensor imaging (DTI) at 3 Tesla and high resolution anatomical images at 7 Tesla, we will detect structural changes in patients with primary focal dystonia in comparison with control subjects. VBM and DTI are methods implemented in the statistical parametric mapping software (SPM2). Magnetic resonance spectroscopy (MRS) will use special software to calculate gamma-aminobutyric acid (GABA) levels in a region of interest.

Outcome measures

VBM and DTI analysis in SPM2 will enable us to make a voxel-wise comparison of local concentration/volume of gray/white matter among these groups of subjects. This study can lead to an improved knowledge of the pathophysiology of primary hand dystonia can help to elucidate dystonia s pathogenesis/etiology and may lead to specific preventative or therapeutic approaches. The MRS study will enable us to study GABA levels in the sensory motor cortices, prefrontal cortex and basal ganglia in primary dystonia patients and normal subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

HEALTHY VOLUNTEERS: Healthy volunteers who consented to participate in the study and matched for age, sex, handedness with the group of patients with primary focal hand dystonia.

PATIENTS: Patient with primary focal dystonia from our dystonia patient database who consented to participate in the study. This criterion will be established by the preliminary screening in the Human Motor Control Outpatient Clinic.

EXCLUSION CRITERIA:

The following subjects will be excluded:

Healthy volunteers with cognitive complaints, abnormal neurological exam or history of past neurological disease.

Dystonia patients with the presence of a second neurological disease or condition; abnormal neurological findings on exam that are not related to primary focal dystonia.

Subjects with past or present neuropsychiatric illness, head trauma with loss of consciousness, epilepsy, cerebro-vascular disease, migraine, past and present history of alcohol abuse, medical conditions that may alter cerebral structure.

Subjects with abnormal MRI findings at visual inspection (prominent normal variants such as mega cisterna or cavum septum pellucidum, signs of severe cortical or subcortical atrophy, brain tumors, vascular diseases, trauma or AVMs).

Subjects with any metallic objects within them just prior to MR imaging (cardiac or neural pacemaker, aneurysm clips [metal clips on the wall of a large artery], metallic prostheses [including heart valves and cochlear implants] or shrapnel fragments. Welders and metal workers are also at risk for injury and may not take part in the study because of possible small metal fragments in the eye of which they may be unaware.

Subjects not capable of giving an informed consent.

Women who are pregnant

Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2002-02-27; Study Completion 2015-03-10

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Berardelli A, Rothwell JC, Hallett M, Thompson PD, Manfredi M, Marsden CD. The pathophysiology of primary dystonia. Brain. 1998 Jul;121 ( Pt 7):1195-212. doi: 10.1093/brain/121.7.1195. PMID 9679773
- [Background] Bhatia KP, Marsden CD. The behavioural and motor consequences of focal lesions of the basal ganglia in man. Brain. 1994 Aug;117 ( Pt 4):859-76. doi: 10.1093/brain/117.4.859. PMID 7922471
- [Background] Lee MS, Marsden CD. Movement disorders following lesions of the thalamus or subthalamic region. Mov Disord. 1994 Sep;9(5):493-507. doi: 10.1002/mds.870090502. PMID 7990845